CLINICAL TRIAL: NCT04571437
Title: Letrozole With or Without Metronomic Capecitabine in First Line Treatment of Patients With ER-positive HER2 Negative Advanced Breast Cancer: A Randomized Phase II Study.
Brief Title: Letrozole and Metronomic Capecitabine in ER-positive HER2 Negative Advanced Breast Cancer (B-001 Study)
Acronym: B-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Saleh, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-127-2019
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Estrogen Receptor-positive Breast Cancer; Metastatic Breast Cancer
Keywords: Advanced breast cancer; chemo-hormonal; hormone positive; metronomic capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Letrozole

STUDY DESIGN:
Intervention Model Description: Patients are assigned into two arms of treatment, arm A contains Letrozole and metronomic Capecitabine while arm B contains Letrozole alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemo endocrine treatment (A) (Active Comparator): Letrozole 2.5mg PO daily + Capecitabine 500mg/m2 bid PO continously
  Interventions: Drug: Capecitabine; Drug: Letrozole 2.5mg
- Endocrine treatment only (B) (Active Comparator): Letrozole 2.5mg PO daily
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Capecitabine — Capecitabine metronomic combined with Letrozole
  Other Names: Xeloda
  Arms: Chemo endocrine treatment (A)
Drug: Letrozole 2.5mg — Letrozole daily alone
  Other Names: Femara

SUMMARY:
A phase II clinical trial designed to test the effect of combining endocrinal therapy (Letrozole) with chemotherapy (Capecitabine) in first line treatment of advanced cases of female breast cancer with ER positive disease.

DETAILED DESCRIPTION:
This is a randomized clinical trial that assigns patients with female breast cancer in the metastatic entity or advanced -beyond local disease treatment - entity into two arms. Arm A contains Letrozole with metronomic Capecitabine versus arm B that contains Letrozole alone. This is to be applied on ER positive HER2 negative tumours.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 18-70
* ECOG-PS 0-II.
* Histopathological proof of breast cancer
* ER positive (Allred score of ≥3 out of 8), and HER2 negative by IHC (or ISH if HER2 +2).
* Metastatic/recurrent disease as proven by CT scan, bone scan or clinical examination (for skin lesions). Biopsy of the recurrent lesions is encouraged but not mandatory.
* Either hormone sensitive setting (Denovo metastatic disease or disease progression after more than 1 year of ending adjuvant endocrine therapy) or secondary resistance to tamoxifen therapy (disease relapse after more than 2 years of starting and less than 1 year of ending adjuvant endocrine therapy, or DP of metastatic disease after more than 6 months of first line tamoxifen).
* Adequate organ function.
* Signed informed consent

Exclusion criteria:

* Inadequate organ functions.
* Disease progression while on prior aromatase inhibitor therapy.
* Primary endocrine resistance.
* Double primary cancer (history of other malignancy apart from a non melanoma skin cancer).
* Refusal to sign consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 204 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
6 months Progression free survival rate | 6 months from the start of treatment
  Percentage of patients alive and progression-free at 6 months

SECONDARY OUTCOMES:
Overall response rate | 6 months from the start of treatment
  Rate of CR+PR as assessed by the investigator using RECIST 1.1 criteria
Adverse events rates in both groups | 6 months from the start of treatment
  Rates of all grade (grade 1-4) and high grade (grade 3+4) adverse events as assessed by NCI-CTAE v4.0
Quality of life assessment using FACIT-B questionnare | 6 months
  FACIT-B questionnare will be completed by each patient at baseline and 6 months after randomization
Median progression free survival | 18 months
  comparison of estimated median PFS between both groups
Time to treatment failure | 18 months
  Time from start treatment to progression, death or treatment discontinuation from any cause
Clinical benefit rate | After 6 months of treatment
  Complete response + partial response + stable disease for 6 months
Overall survival | 24 months
  Percentage of patients alive at 24 months
Time to chemotherapy adminstration | 18 months
  Time from randomization to the first chemotherapy administration

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Saleh, M.D, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azim HA, Saleh MA, Essam Eldin P, Abdelhafeez AAM, Hassan M, Kassem L. Combination of metronomic capecitabine and letrozole in metastatic hormone receptor positive, HER2 negative breast cancer: a randomized phase II trial. J Chemother. 2025 Apr;37(2):159-167. doi: 10.1080/1120009X.2024.2342741. Epub 2024 May 20. PMID 38764430